CLINICAL TRIAL: NCT02907112
Title: Impact of Reducing Dietary Intake of Red and Processed Meat Intake on Fasting Lipemia in Healthy Participants
Acronym: ELM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TS/L005891/1
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Lipidemia
Keywords: meat intake; meat analogues; LDL Cholesterol; HDL Cholesterol
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participants to continue on their habitual diet for 4 weeks
- Meat Reduction (Experimental): Participants asked to reduce their red and processed meat intake by 50% for 12 weeks
  Interventions: Behavioral: Meat reduction

INTERVENTIONS:
Behavioral: Meat reduction — Advice, Motivational material and food products provided to participants
  Arms: Meat Reduction

SUMMARY:
Excessive meat consumption, particularly of red and processed meat, is associated with increased risk of developing a range of chronic diseases. Meat production also significantly contributes to the production of global greenhouse gasses (GHG). Given the predicted global increase in the human population, coupled with the rise in demand for meat within emerging economies, it has been suggested that strategies to alter dietary patterns and reduce meat intake should be devised. With the provision of appropriate non- or reduced-meat alternatives, this study aims to investigate whether free living subjects can significantly reduce their meat intake, and whether such dietary changes positively impact on a range of health measures

DETAILED DESCRIPTION:
In UK adults, meat provides approximately 40% of the average daily protein intake and makes a significant contribution to intake of thiamin, niacin, vitamin B12, iron, zinc, potassium, and phosphorus. However, excessive consumption, particularly of red and processed meat, is associated with increased risk of developing a range of chronic diseases, including cardiovascular disease (CVD), obesity, type 2 diabetes and some cancers. Meat production significantly contributes to the production of greenhouse gasses (GHG) and hence global warming. Given the predicted global increase in the human population, coupled with the rise in demand for meat within emerging economies, it has been suggested that concerted efforts should be made to alter dietary patterns and reduce meat intake. Moreover, a number of reports have suggested that replacing meat with non-meat protein-rich products has health benefits. Such products tend to be inherently lower in total and saturated fat and, higher in fibre and as such, could also be cardioprotective.

The aim of this trial will be to investigate whether, with appropriate non/reduced-meat alternatives and motivational support, free living subjects can significantly reduce their meat intake and whether such dietary changes positively impact on a range of cardiovascular risk factors.

Trial design; A non-randomised, single group study design, with an initial control period will be used.

Participants; Forty healthy men and women will be recruited from the general population of Nottinghamshire, UK. All participants will attend the David Greenfield Human Physiology Unit (Queen's Medical Centre, Nottingham, UK) for an initial medical screening visit to confirm health status. In addition, blood pressure (BP) will be measured at the left upper arm (after lying semi-supine for 5min) using automated oscillometry, and body mass index (BMI) will be calculated from measured height and weight. If participants are suitable to take part with regards to their health questionnaire and BMI measures, a venous blood sample will then be taken to assess full blood count, urea, and electrolytes. Those taking lipid-lowering medication, or who report using nutritional strategies to lower their cholesterol, will be excluded. Participants will be accepted onto the trial if they report habitual consumption of 4-5 portions of red and/or processed meat per week (with 3-4 of these being consumed as main meals), they do not have food allergies related to soya or mycoprotein, and do not demonstrate any clinically significant abnormalities on screening.

Study Protocol; After recruitment, participants will be asked to record all food intake (including snacks and drinks) in a diet diary, for 4 days (3x week or work days, and 1x weekend or rest day) prior to assessment visit 1, for baseline assessment of macronutrient and energy intake. Individuals will be asked to complete further 4-day diet diaries in the week before assessment visits 2,3 and 4 (weeks 4, 10, and 16), to assess any changes in macronutrient or energy intake and meat consumption which may have occurred as a consequence of the intervention. Household measures will be used to estimate portion size, and diaries will be analysed using a food composition database. To calculate habitual diet composition, a mean daily intake will obtained from all 4 days of each recording period, and these data will be combined to produce group means.

Assessment visits will take place in the morning after the individual has fasted from midnight the night before. Initially, measurement of body mass will be made to the nearest 0.1kg using a Seca 882 Digital Scale, and waist and hip circumference will be assessed (with the participant standing) mid-way between the lowest rib and the iliac crest, and at the greater trochanters, respectively. Participants will then be asked to rest, semi-supine, on a couch for >5min before having their resting BP measured, and estimation of body composition made using bioelectrical impedance. A 5ml fasting blood sample will be taken for determination of serum insulin, total cholesterol, high density lipoprotein cholesterol (HDL), low density lipoprotein cholesterol (LDL), triacyl glycerides (TAG) and whole blood glucose. In a subset of the cohort (n=26, 13 Male:13 Female), flow mediated dilatation (FMD) will also be measured on the laboratory visits when fasted, after resting semi-supine for 1 and 2 hours.

Intervention; After visit 1 (week 0) assessment, participants will be asked not to make any changes to their lifestyle and to continue their habitual diet until visit 2 (week 4) when a second assessment will be made ('control' period). The 12 week 'intervention' period will begin on the day after the second study visit. Participants will be given information regarding how meat intake can safely be reduced in their diet, including a recipe book containing ideas for meals using meat analogues and other protein sources. A range of frozen meat-free (soya or mycoprotein 'mince', mycoprotein sausages, meatballs and 'steak strips') and reduced meat products (pork sausages, beef meatballs, beef mince and beef burgers made with 50% meat and 50% soya or mycoprotein) are available for the participants to use to aid this reduction in red meat intake. In addition, a range of dried beans (red kidney, haricot, black turtle), pulses (chick peas, green and red lentils) and grains (quinoa) will also be offered. Weekly telephone contact with the study participants will be maintained over the intervention period to improve compliance, to identify any problems and to arrange further food deliveries.

ELIGIBILITY:
Inclusion Criteria:

BMI 18 - 28 kg/m2 Healthy Females should be premenopausal Good spoken and written English Consume 4-5 portions of red and/or processed meat per week consumption of greater than 70g per day

Exclusion Criteria:

Smoking Chronic diseases Hypertension Pregnancy / Breast feeding Chronic medication use (excluding oral contraceptives) Participation in any other research study three months prior to the screening or during study duration Clinically significant findings at screening

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Fasting Serum total cholesterol concentration | Week 0, 4,10 and 16
  Fasting Serum total cholesterol concentration

SECONDARY OUTCOMES:
Fasting Serum LDL cholesterol concentration | Week 0, 4,10 and 16
  Fasting Serum LDL cholesterol concentration
Fasting Serum HDL cholesterol concentration | Week 0, 4,10 and 16
  Fasting Serum HDL cholesterol concentration
Fasting whole blood glucose concentration | Week 0, 4,10 and 16
  Fasting whole blood glucose concentration
Fasting Serum Insulin concentration | Week 0, 4,10 and 16
  Fasting Serum Insulin concentration
Resting, supine blood pressure | Week 0, 4,10 and 16
  Resting, supine blood pressure (systolic and diastolic)
Body mass index calculated from measured height and weight (BMI) | Week 0, 4,10 and 16
  Body mass index calculated from measured height and weight (BMI)
% body fat determined by Bio-electrical Impedance | Week 0, 4,10 and 16
  % body fat determined by Bio-electrical Impedance
Flow-mediated dilatation | Week 0, 4 and 16
  Flow mediated dilatation at the brachial artery, measured using ultrasound (in a subset of participants)
Quality of Life Questionnaire | Week 0, 4,10 and 16
  WHOQOL Questionnaire
Dietary macro-nutrient intake | Week 0, 4,10 and 16
  Macro-nutrient intake of the diet determined from diet diaries
Dietary energy intake | Week 0, 4,10 and 16
  Energy intake of the diet determined from diet diaries
Meat intake | Week 0, 4,10 and 16
  daily red and processed meat intake determined from diet diaries
Full blood count | Week 0,10 and 16
  blood cell count, including haemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Salter, PhD, Principal Investigator — University of Nottingham
Locations (1):
- David Greenfield Human Physiology Unit, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Simpson EJ , Clark M , Razak AA , Salter A . The impact of reduced red and processed meat consumption on cardiovascular risk factors; an intervention trial in healthy volunteers. Food Funct. 2019 Oct 16;10(10):6690-6698. doi: 10.1039/c9fo00758j. PMID 31559410